CLINICAL TRIAL: NCT07336901
Title: Comparison of Adductor Canal Block and IPACK Block Versus Adductor Canal Block and the Gastrosoleus Interfascial Plane Block for Postoperative Analgesia After Total Knee Arthroplasty: a Prospective Double Blinded Study
Brief Title: Adductor Canal Block and IPACK Block vs Adductor Canal Block and the Gastrosoleus Interfascial Block After Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, alyaa abdel sattar mohamed hassan, lecturer, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R761
Record Dates: First submitted 2025-12-26; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Pain After Knee Arthroplasty
Keywords: gastrosoleus interfascial plane block, knee arthroplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACB/GIP group (Experimental): Adductor canal block will be given. In supine position, the leg will be externally rotated and the probe will be positioned at the midpoint of the thigh on its medial aspect. The adductor canal (AC) will be located anterolaterally to the superficial femoral artery deep to the sartorius muscle. The needle (size) will be advanced and a particular "pop" will be felt when the tip pierced the vastoadductor membrane, which is the roof of the adductor canal. A single dose of (20 ml of 0.25% bupivacaine) will be injected.
  The gastrosoleus interfascial plane block will be given along the medial border of the leg in long axis, 7 cm-8 cm below the popliteal crease. After identification of muscle bellies of the medial gastrocnemius head, the soleus and the trilaminar fascial plane between these muscles, 20 ml of bupivacaine 0.25% will be injected at this plane by piercing the fascia.
  Interventions: Procedure: Adductor Canal Block (ACB) + gastrosoleus interfascial plane block
- ACB/IPACK group (Experimental): Adductor canal block will be given. In supine position, the leg will be externally rotated and the probe will be positioned at the midpoint of the thigh on its medial aspect. The adductor canal (AC) will be located anterolaterally to the superficial femoral artery deep to the sartorius muscle. The needle (size) will be advanced and a particular "pop" will be felt when the tip pierced the vastoadductor membrane, which is the roof of the adductor canal. A single dose of (20 ml of 0.25% bupivacaine) will be injected.
  The patients will receive IPACK with the patient placed in a supine position and knee placed in position of 90° flexion. By placing a low-frequency ultrasound probe in the popliteal crease the spinal needle will be advanced from medial aspect of the knee going from anteromedial to posterolateral between the popliteal artery and the femur. The tip of the needle will be placed 1-2 cm beyond the lateral edge of the artery, and 20 ml of 0.25% bupivacaine will be injected.
  Interventions: Procedure: Adductor Canal Block (ACB) + iPACK Block

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) + gastrosoleus interfascial plane block — Adductor canal block will be given. In supine position, the leg will be externally rotated and the probe will be positioned at the midpoint of the thigh on its medial aspect. The adductor canal (AC) will be located anterolaterally to the superficial femoral artery deep to the sartorius muscle. The needle (size) will be advanced and a particular "pop" will be felt when the tip pierced the vastoadductor membrane, which is the roof of the adductor canal. A single dose of (20 ml of 0.25% bupivacaine) will be injected.
  The patients will receive gastrosoleus interfascial plane block. Using a linear probe the transducer will be placed along the medial border of the leg in long axis, 7 cm-8 cm below the popliteal crease. After identification of muscle bellies of the medial gastrocnemius head, the soleus and the trilaminar fascial plane between these muscles, 20 ml of bupivacaine 0.25% will be injected at this plane by piercing the fascia (loss of resistance).
  Arms: ACB/GIP group
Procedure: Adductor Canal Block (ACB) + iPACK Block — Adductor canal block will be given. In supine position, the leg will be externally rotated and the probe will be positioned at the midpoint of the thigh on its medial aspect. The adductor canal (AC) will be located anterolaterally to the superficial femoral artery deep to the sartorius muscle. The needle (size) will be advanced and a particular "pop" will be felt when the tip pierced the vastoadductor membrane, which is the roof of the adductor canal. A single dose of (20 ml of 0.25% bupivacaine) will be injected.
  The patients will recieve IPACK with the patient placed in a supine position and knee placed in position of 90° flexion. By placing a low-frequency ultrasound probe in the popliteal crease the spinal needle will be advanced from medial aspect of the knee going from anteromedial to posterolateral between the popliteal artery and the femur. The tip of the needle will be placed 1-2 cm beyond the lateral edge of the artery, and 20 ml of 0.25% bupivacaine will be injected.
  Arms: ACB/IPACK group

SUMMARY:
Evaluate analgesic efficacy of adductor canal block with IPACK versus that of adductor canal block with gastrosoleus interfascial plane block in total knee arthroplasty surgeries.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a surgical procedure commonly known for its association with sever postoperative pain. This pain can affect quality of recovery by restricting patient's ability to mobilize early and participate effectively in rehabilitation, which eventually will prolong hospital stays and increase healthcare costs. Also chronic postsurgical pain may complicate inadequately managed postsurgical pain.

Hence the need for exploring different analgesic modalities has evolved involving different techniques either regional anesthesia or systemic analgesics.

Peripheral nerve blockade was found to achieve adequate postoperative pain relief, and techniques such as sciatic nerve block, femoral nerve block and adductor canal block have been introduced.

Adductor canal block (ACB) has been shown to decrease pain significantly and thereby opioid consumption with minimal effect on quadriceps function.

Though ACB provides analgesia to the peripatellar and intra-articular aspect of knee joint, it does not relieve posterior knee pain which may compromise satisfactory pain relief.

Infiltration of the interspace between popliteal artery and the capsule of posterior knee (IPACK) by local anesthetics has been achieved by ultrasound and was found to provide significant posterior knee analgesia. Its technique was described by Elliott et al.

Recently the gastrosoleus interfascial plane block (GIP) was introduced in 2023 by Abraham et al which targets the fascial plane between the soleus muscle and the medial belly of the gastrocnemius muscle.

All patients will be preoperatively assessed then connected to basic monitors (ECG, NIBP and SpO2) IV line will be inserted and crystalloid fluid infusion will be started Patients will be premedicated by midazolam (1-2 mg), and they will be pre oxygenated 3-5 minutes before induction of anesthesia. General anesthesia will be given using propofol 2-3mg/kg intravenous (IV), fentanyl 1-2µg/kg IV and atracurium 0.5 mg/kg IV as a muscle relaxant to facilitate intubation. Anesthesia will be maintained by isoflurane and atracurium 0.1-0.2 mg/kg every 20-30 minutes. Patients will be mechanically ventilated with 50% O2 and 50% air keeping end-tidal CO2 between 30 - 35 mmHg. Fentanyl bolus doses of 0.5-1 mcg/kg will be given according to the changes of hemodynamic variables (more than 20% base line).

Adductor canal block will be given to both groups. In supine position, the leg will be externally rotated and the probe will be positioned at the midpoint of the thigh on its medial aspect. The adductor canal (AC) will be located anterolaterally to the superficial femoral artery deep to the sartorius muscle. The needle (size) will be advanced and a particular "pop" will be felt when the tip pierced the vastoadductor membrane, which is the roof of the adductor canal. A single dose of (20 ml of 0.25% bupivacaine) will be injected.

The patients in group A will receive gastrosoleus interfascial plane block. The patients in Group B will receive IPACK with the patient placed in a supine position and knee placed in position of 90° flexion At PACU, all patients will receive paracetamol 1gm to be repeated every 8 hours.

Patients' pain will be assessed using VAS score (12) in the PACU and every 4 hours thereafter for two days. Patient with VAS score ≥4 will recieve a rescue dose of morphine 3-5 mg.

Vital signs including heart rate, systolic and diastolic BP, and oxygen saturation will be recorded intra operatively every 15 min and postoperatively every 4 hours while assessing pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA class I to III of both sexes
* undergoing unilateral total knee arthroplasty
* 40-80 years old

Exclusion Criteria:

* Patient refusal
* History of coagulopathies
* Severe renal insufficiency
* Preexisting lower limb neurological abnormality
* Known allergic history to any of the drugs used in this study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain using visual analogue score VAS score | change in VAS score 30 min after arrival to PACU change in VAS score 4 hours after arrival to PACU change in VAS score 8 hours after arrival to PACU change in VAS score 12 hours after arrival to PACU change in VAS score 24 hours after arrival to PACU
  • Postoperative pain using vas score where 0 is worst pain, 10 is no pain

SECONDARY OUTCOMES:
Time to first morphine analgesic dose and total rescue doses of morphine. | time needed for patient to use morphine in hours after end of surgery
  Time to first morphine analgesic dose in hours.
cumulative doses of morphine | cumulative doses of morphine in mg in the first 24 hours after operation
  cumulative doses of morphine in mg
Range of motion by assessing degree of knee extension 24 hours after surgery. | Assessing degree of knee extension 24 hours after surgery.
  Range of motion by assessing degree of knee extension 24 hours after surgery.
Time of first postoperative ambulation and how many feets the patient will be able to walk. | Time of first postoperative ambulation and how many feets the patient will be able to walk in the 24 hours after operation
  Time of first postoperative ambulation and how many feets the patient will be able to walk.
Duration of postoperative hospital stay. | Duration of postoperative hospital stay in days
  Duration of postoperative hospital stay.
complications of the block | complications of the block (vascular injury, nerve injury, allergic reaction) in the 24 hours after surgery
  vascular injury, nerve injury, allergic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Alyaa A Hassan, lecturer, Principal Investigator — Faculty of medicine, Fayoum university; Mohamed A Shawky, Associate professor, Study Director — Faculty of medicine, Fayoum university; Omar S Farghaly, Associate professor, Principal Investigator — Faculty of medicine, Fayoum university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korean Knee Society. Guidelines for the management of postoperative pain after total knee arthroplasty. Knee Surg Relat Res. 2012 Dec;24(4):201-7. doi: 10.5792/ksrr.2012.24.4.201. Epub 2012 Nov 29. PMID 23269957
- [Background] Kim DH, Pearson-Chauhan KM, McCarthy RJ, Buvanendran A. Predictive Factors for Developing Chronic Pain After Total Knee Arthroplasty. J Arthroplasty. 2018 Nov;33(11):3372-3378. doi: 10.1016/j.arth.2018.07.028. Epub 2018 Aug 4. PMID 30143334